CLINICAL TRIAL: NCT02014740
Title: Effect of Liraglutide on Epicardial Fat in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Gianluca Iacobellis, Professor of Clinical Medicine, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20120811
Record Dates: First submitted 2013-12-12; First posted 2013-12-18 (Estimated); Results first posted 2018-03-22 (Actual); Last update posted 2019-06-06 (Actual); Status verified 2019-06

CONDITIONS: Type 2 Diabetes; Overweight; Obesity
Keywords: Epicardial fat; Type 2 diabetes; Obesity; GLP-1 analogs
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Overweight; Obesity | interventions — Liraglutide; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Liraglutide (Experimental): • L-group will be started and dose-escalated to 1.8mg sc once daily according to below schedule: Liraglutide will be administered with a starting dose of 0.6 mg (after a least one week) and subsequent increments to 1.2 mg (after a least one week) and to 1.8 mg (after at least a week on 1.2 mg). L-group subjects will need to achieve the final dose of 1.8 mg by at least three weeks from the starting dose. Subjects who would not be able to achieve the dose of 1.8 mg (due to potential side effects) will be advised to lower the dose to 1.2 mg. Metformin regimen will be continued.
  Interventions: Drug: Liraglutide; Drug: Metformin
- Metformin (Active Comparator): M-group will be treated with Metformin for the duration of the study. Metformin (from 500 mg twice daily to a maximum of 1000 mg twice daily) regimen will be continued to achieve fasting glucose between 80 and 140 mg/dl
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Liraglutide — Liraglutide (Victoza) is an acylated analogue of glucagon-like peptide-1 (GLP-1) indicated for the treatment of type 2 diabetes mellitus• L-group will be started and dose-escalated to 1.8mg sc once daily according to below schedule: Liraglutide will be administered with a starting dose of 0.6 mg (after a least one week) and subsequent increments to 1.2 mg (after a least one week) and to 1.8 mg (after at least a week on 1.2 mg). L-group subjects will need to achieve the final dose of 1.8 mg by at least three weeks from the starting dose. Subjects who would not be able to achieve the dose of 1.8 mg (due to potential side effects) will be advised to lower the dose to 1.2 mg. Metformin regimen will be continued. .
  Arms: Liraglutide
Drug: Metformin

SUMMARY:
The purpose of this research study is to learn about the effect of Liraglutide, (Victoza®), on the fat surrounding the heart.Excessive amount of the fat around the heart is common in people with type 2 diabetes and can be associated with poor sugar control. Liraglutide is an injectable prescription medicine that can improve blood sugar control in adults with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes, as defined by ADA criteria
* HbA1c < 8% measured at least 1 month prior to this study
* BMI ≥27 kg/m2
* Pre-treatment with Metformin
* Age > 18 and < 65 years old

Exclusion Criteria:

* • Known contra-indications to Liraglutide, such as previous history of pancreatitis or medullary thyroid carcinoma, personal or family history of MEN, in accordance with risks and safety information included in the latest updated Prescribing Information for Victoza®

  * Type 1 diabetes, as defined by American Diabetes Association (ADA) criteria
  * Insulin dependent or treated type 2 diabetes
  * Current use of other injectable incretins
  * History of diabetes ketoacidosis
  * Advanced Chronic Kidney Disease, as defined by Glomerular Filtration Rate (GFR) < 30 mL/min/1.73m2
  * Clinical signs or symptoms of New York Heart Association (NYHA) class III-IV heart failure
  * Clinical or laboratory evidences of chronic active liver diseases
  * Acute or chronic infective diseases
  * Cancer or chemotherapy
  * Current use of systemic corticosteroids or in the 3 months prior this study
  * Known or suspected allergy to Liraglutide, excipients, or related products
  * Pregnant, breast-feeding or the intention of becoming pregnant
  * Females of childbearing potential who are not using adequate contraceptive methods

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-03; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Miami, Miami, Florida, United States

REFERENCES:
- [Derived] Iacobellis G, Mohseni M, Bianco SD, Banga PK. Liraglutide causes large and rapid epicardial fat reduction. Obesity (Silver Spring). 2017 Feb;25(2):311-316. doi: 10.1002/oby.21718. PMID 28124506

RESULTS

PARTICIPANT FLOW:
Groups:
- Liraglutide: L-group will be started and dose-escalated to 1.8mg sc once daily according to below schedule: Liraglutide will be administered with a starting dose of 0.6 mg (after a least one week) and subsequent increments to 1.2 mg (after a least one week) and to 1.8 mg (after at least a week on 1.2 mg). L-group subjects will need to achieve the final dose of 1.8 mg by at least three weeks from the starting dose. Subjects who would not be able to achieve the dose of 1.8 mg (due to potential side effects) will be advised to lower the dose to 1.2 mg. Metformin regimen will be continued.
- Metformin: M-group will be treated with Metformin for the duration of the study. Metformin (from 500 mg twice daily to a maximum of 1000 mg twice daily) regimen will be continued to achieve fasting glucose between 80 and 140 mg/dl
  Metformin
Period: Overall Study
Arm/Group | Liraglutide | Metformin
Started | 55 | 45
Completed | 49 | 40
Not Completed | 6 | 5
Not completed — Lost to Follow-up | 4 | 4
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Liraglutide | Metformin | Total
Number analyzed (Participants) | 55 | 45 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 55 | 45 | 100
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (10) | 52 (10) | 50.8 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 28 | 61
  Male | 22 | 17 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21 | 17 | 38
  Not Hispanic or Latino | 34 | 28 | 62
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 55 | 45 | 100
Epicardial adipose tissue Thickness (EAT) [Mean (Standard Deviation); unit: mm] | 9.6 (2) | 7.4 (1.6) | 8.75 (1.9)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 37.8 (7) | 32.6 (6) | 35.2 (6)
HemoglobinA1c (HbA1c) [Mean (Standard Deviation); unit: %] | 6.6 (0.8) | 6.4 (0.6) | 6.52 (0.6)

OUTCOME MEASURES:

1. Primary Outcome: Echocardiographic Epicardial Fat Thickness
Description: Echocardiographic epicardial fat thickness is an non invasive, inexpensive, reproducible and direct measure of visceral fat. In fact, epicardial fat strongly reflects the intra-abdominal and intra-myocardial fat accumulation as measured by magnetic resonance imaging procedures.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Liraglutide | Metformin
Number analyzed (Participants) | 55 | 45
mm
  Baseline | 9.6 (2) | 7.4 (1.6)
  3-month | 6.8 (1.5) | 7.5 (1.5)
  6-month | 6.2 (1.5) | 6.9 (1.5)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Liraglutide | Metformin
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/45
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/45
Other Adverse Events (participants affected / at risk) | 16/55 | 12/45
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Liraglutide (N=55) | Metformin (N=45)
nausea (Gastrointestinal disorders) | 16 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-12-05): https://cdn.clinicaltrials.gov/large-docs/40/NCT02014740/Prot_SAP_ICF_000.pdf